CLINICAL TRIAL: NCT04731051
Title: A Pilot, Randomized, Open-label Trial to Determine the Feasibility, Safety, Efficacy, and Pharmacokinetics of Nebulized HCQ01 for the Treatment of Patients With COVID-19 and Cancer
Brief Title: The Potential Use of Inhaled Hydroxychloroquine for the Treatment of COVID-19 in Cancer Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: the study was terminated as no more COVID cases were treated at the center
Sponsor: King Hussein Cancer Center (Other)
Collaborators: Amman Pharmaceutical Industries (API) (Unknown); Sana Pharmaceutical Industry (Unknown); ACDIMA Biocenter (Other)
Responsible Party: Principal Investigator, Feras Hawari, Consultant in Pulmonary and Critical Care, King Hussein Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYDR0121/CCO
Record Dates: First submitted 2021-01-28; First posted 2021-01-29 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: 2019 Novel Coronavirus
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Arm (Hydroxychloroquine sulfate, 5 days) (Experimental): Participants will receive continued standard of care therapy (SOC) for COVID-19 together with 2 ml HCQ01 (12.5 mg/ml) twice a day for 5 consecutive days.
  Interventions: Drug: HCQ01; Drug: standard of care (SOC) for COVID-19
- Second Arm (Continued Standard of Care (SOC) Therapy) (Active Comparator): Participants will receive continued standard of care therapy for COVID-19
  Interventions: Drug: standard of care (SOC) for COVID-19

INTERVENTIONS:
Drug: HCQ01 — HCQ01 is a sterile, clear and colorless, ready-to-use aqueous nebulizer solution. Hydroxychloroquine sulfate administered via nebulization
  Arms: First Arm (Hydroxychloroquine sulfate, 5 days)
Drug: standard of care (SOC) for COVID-19 — Standard of care (SOC) for COVID-19

SUMMARY:
This is a pilot, randomized, single-center, parallel group, open-label controlled study to evaluate the feasibility, safety, efficacy, and pharmacokinetics of nebulized HCQ01 plus Standard of Care (SOC) versus SOC alone in hospitalized cancer patients with COVID-19. King Hussein Cancer Center (KHCC) is the study sponsor, and the study will be conducted at KHCC COVID-19 wards.

Approximately 28 cancer patients, ≥18 years of age with a confirmed SARS-CoV-2 infection, will be enrolled and randomized 1:1 to the treatment and control arms where they will receive ten doses of Hydroxychloroquine solution via nebulizer in addition to SOC or the control arm where treatment will follow KHCC SOC.

ELIGIBILITY:
Inclusion criteria:

1. Documented informed consent of the patient and/or legally authorized representative. Assent, when appropriate, will be obtained per institutional guidelines.
2. Male or female ≥18 years of age at time of enrolment.
3. History of/ or active histologically or cytologically confirmed diagnosis of hematological or solid tumor (any type, any stage and any localization).
4. Eastern Cooperative Oncology Group (ECOG) Status < or = 3 (Appendix I).
5. Patients must have an active cancer treatment or have completed therapy within 12 months of initiation of protocol specified therapy. This includes:

   * Patients with a new cancer diagnosis who have not yet initiated cancer therapy.
   * Patients on active or have recently completed cancer-directed therapy including chemotherapy, targeted therapy, radiation therapy, immunotherapy or hormonal therapy amongst others which would not increase the risk of having an adverse outcome from participating in this study.
6. Currently hospitalized with laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) collected within one week prior to randomization.
7. Initial COVID-19 severity status on the WHO 11-point Ordinal Scale for Clinical Improvement = 4 ("Hospitalized; no oxygen therapy "), = 5 ("Hospitalized; oxygen by mask or nasal prongs "), or 6 ("Hospitalized; oxygen by NIV or high flow ") (Appendix II).
8. COVID-19-induced pneumonia evidenced by chest X-ray, computed tomography scan (CT scan) or magnetic resonance scan (MR scan).
9. Estimated life expectancy of at least 6 months at hospital admission for COVID-19.
10. Patients must be receiving standard of care for SARS-CoV-2.
11. Patients must have an assessment of adequate organ function within 28 days prior to enrolment, evidenced by:

    * Hemoglobin ≥ 9.0 g / dL.
    * Leukometry> 2,000 / mm3 (> 2 10E3/ ul).
    * Absolute neutrophil count ≥ 1,500 / mm3 (≥1.5 10E3/ul).
    * Platelet count ≥ 100,000 / mm3 (≥100 10E3/ul).
    * Creatinine clearance ≥ 30 mL / min. Creatinine clearance (CrCl) should be calculated according to the Cockcroft-Gault formula.
    * Total bilirubin <3 x the upper limit of normal (ULN), except for patients with known Gilbert's syndrome.
    * Aspartate aminotransaminase (AST) <3.0 x LSN.
    * Alanine aminotransaminase (ALT) <3.0 x ULN.

Exclusion criteria:

1. Pregnant (positive β-human chorionic gonadotropin test, β-HCG) or lactating female at screening.
2. Patients with a history of retinopathy, sickle cell disease or trait, psoriasis, porphyria, history of splenectomy, mental illness or uncontrolled seizures disorder, known active tuberculosis or history of incompletely treated tuberculosis, patients on chronic immunosuppression for other medical conditions such as rheumatological disorders, inflammatory bowel disease, or in patients with organ transplants.
3. Patients admitted in ICU.
4. Taking medications which may lead to interactions with hydroxychloroquine, including penicillamine, telbivudine, botulinum toxin, fluconazole, digoxin, propafenone , cimetidine, statins, warfarin, and cyclosporine within 2 weeks of dosing start, and during the duration of the study.
5. History of Glucose-6-phosphate dehydrogenase deficiency.
6. Pre-treatment corrected QT interval (QTc) ≥450 milliseconds.
7. Acute or chronic kidney disease (stage-4 or -5 renal impairment; eGFR<30 mL/min/1.73 m2 or hemodialysis).
8. Liver Child-Pugh grade C.
9. Patients with Hypokalemia (<3.6 mg/dl), Hypocalcemia (<8.8 mg/dl), Hypomagnesemia (<1.7 mg/dl). Will be included after correction.
10. Need for mechanical ventilation.
11. History of hypersensitivity to hydroxychloroquine.
12. History of Chronic Hepatitis B or hepatitis C infections.
13. History of Human Immunodeficiency Virus (HIV) infection.
14. Concurrent serious illness including, but not limited to, any of the following:

    * Clinically significant cardiovascular disease (e.g., uncontrolled hypertension, myocardial infarction, or unstable angina).
    * New York Heart Association class II-IV congestive heart failure.
    * Serious cardiac arrhythmia requiring medication.
    * Peripheral vascular disease ≥ grade 2 within the past year.
    * Psychiatric illness/social situation that would limit compliance with study requirements.
    * COPD, Lung cancer, and moderate to severe asthma.
15. Any other significant finding based on the judgment of the PI would increase the risk of having an adverse outcome from participating in this study.
16. Any other concomitant treatment based on the judgment of the PI would increase the risk of having an adverse outcome from participating in this study.
17. Is currently participating in or has participated in an interventional clinical trial with an investigational compound or device within 80 days of signing the informed consent/assent for this current trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who improve by at least one level lower on the 11-point World Health Organization Ordinal Scale for Clinical Improvement (WHO-OSCI), where patients are scored on a scale of 0-10 with 0 being uninfected and 10 being dead . | Time Frame: Day 14

SECONDARY OUTCOMES:
Proportion of participants who improve by at least one level lower on the 11-point WHO-OSCI | Days 5, 28
Change in condition measured using the 11-point WHO-OSCI | Days 5, 14, 28
All-cause mortality | Day 28
Hydroxychloroquine (HCQ) concentration in plasma versus time profiles | Day 1 pre-dose (time 0) and +2, +5, +10, +15, +20, +25, and +30 minutes after dose, and also +1, +2, +3, +4 and +6 hours post-dose completion
Change from Baseline Oxygenation as determined by the SpO2 / FiO2 ratio | Day 5 of treatment
Treatment-related adverse events of HCQ | Up to day 28
  Incidence and severity of treatment-related adverse events.
Rate of Transfer to the Intensive Care Unit | Up to day 28
Time to Clinical Improvement | Up to day 28
  time (in days) to improvement in clinical status by at least one level lower on the 11 point WHO-OSCI
Duration of hospitalization | Up to 28 days
Time to Hospital Discharge OR NEWS2 (National Early Warning Score 2) of ≤ 2 maintained for 24 hrs | Up to 28 days
Status of discharged or not requiring supplemental oxygen | Day 14, 28
Rates of Intensive Care Unit mortality | Day 14, 28
Intensive Care length of stay | Up to day 28
Oxygenation free days | Day 14, 28
Ventilator free days | Day 14, 28
Incidence & duration of new oxygen use | Day 14, 28
Incidence and duration of new mechanical ventilation use | Day 14, 28
Cardiac Arrhythmia - Polymorphic Ventricular Tachycardia | Up to day 28
Cardiac Arrhythmia - Ventricular Tachycardia | Up to day 28
  Cardiologist Diagnostic Documentation
Cardiac Arrhythmia - Lengthening QTc | Up to day 28
  Cardiologist Diagnostic Documentation

CONTACTS AND LOCATIONS:
Overall Officials: Feras Hawari, MD, Principal Investigator — King Hussein Cancer Center
Locations (1):
- King Hussein Cancer Center, Amman, Jordan